CLINICAL TRIAL: NCT04087057
Title: Understanding Barriers Associated With Timely Chemotherapy Administration Among Breast Cancer Patients
Brief Title: Barriers Associated With Timely Adjuvant Chemotherapy Administration in Patients With Invasive Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-1133; NCI-2019-05917 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1133 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Invasive Breast Carcinoma
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (interview, medical records review): Patients complete questionnaires and participate in an interview to answer questions about information patients received before starting chemotherapy, any medical problems after surgery that could have been related to the start of the chemotherapy, how chemotherapy affected patients' life, and anything else patients may remember between the time when the breast surgery ended and the first dose of chemotherapy started. Patients' medical records are also reviewed.
  Interventions: Other: Interview; Other: Medical Chart Review; Behavioral: Questionnaire

INTERVENTIONS:
Other: Interview — Participate in interview
Other: Medical Chart Review — Patients' medical records are reviewed
  Other Names: Chart Review
Behavioral: Questionnaire — Complete questionnaires
  Other Names: Questionnaires

SUMMARY:
This trial studies the barriers associated with timely chemotherapy given after surgery (adjuvant) in patients with invasive breast cancer. Meeting with patients and asking questions may help doctors to learn about factors that can cause delays in the start of chemotherapy after surgery in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To comprehensively and qualitatively assess and identify the determinants of time to chemotherapy (TTC) delays in a vulnerable population using qualitative methods.

Ia. To describe the health literacy/numeracy, social support and level of trust in physicians of the study participants. (Exploratory)

OUTLINE:

Patients complete questionnaires and participate in an interview to answer questions about the information patients received before starting the chemotherapy, any medical problems after the surgery that could have been related to the start of the chemotherapy, how the chemotherapy affected patients' life, and anything else patients may remember between the time when the breast surgery ended and the first dose of chemotherapy started. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary invasive breast cancer
* For patients receiving adjuvant chemotherapy: First dose of chemotherapy administered >= 60 days after definitive breast cancer surgery. For patient treated with neoadjuvant chemotherapy: First dose of chemotherapy administered >= 60 days after pathological diagnosis
* Diagnosis of breast cancer within three years of study enrollment
* Can speak, read, and understand English and/or Spanish
* Patient of Lyndon B. Johnson General Hospital-Harris Health System (LBJ-HHS) or MD Anderson Cancer Center

Exclusion Criteria:

* Women hospitalized for a critical condition or who are considered medically unstable by their medical team
* Patients that started chemotherapy >= 3 years after definitive breast cancer surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Assessment of data collected from individual semi-structured interviews | Up to 1 year
  Will be analyzed using an open code method by identifying and classifying interview data. Qualitative analysis will be done in partnership with a qualitative research consulting group (ResearchTalk, Inc.). Transcripts of the semi-structured interviews will be de-identified by removing 18 protected health information (PHI) identifiers from the transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Chavez Mac Gregor, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org